CLINICAL TRIAL: NCT06803173
Title: Pelvic Floor Muscle Activity in Primary Dysmenorrhea
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wafaa Abdelraouf Mohamed Mohamed, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/005371
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group of mild primary dysmenorrhea: It will consist of 26 females with mild dysmenorrhea (WaLIDD score =1-4)
  Interventions: Other: No intervention
- group of moderate primary dysmenorrhea: It will consist of 26 females with moderate dysmenorrhea (WaLIDD score =5-7)
  Interventions: Other: No intervention
- group of severe primary dysmenorrhea: It will consist of 26 females with severe dysmenorrhea (WaLIDD score =8-12)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study will be conducted to assess the pelvic floor muscle (PFM) activity in primary dysmenorrhea (PD).

DETAILED DESCRIPTION:
Dysmenorrhea, marked by painful menstrual cramps, often involves increased PFM tension, spasms, and inflammation, affecting females' quality of life and productivity. The traditional focus has been on investigating the abdominal region in women with PD. However, this new perspective considers that the hormonal changes experienced during the menstrual cycle in PD patients may lead to a heightened sensitivity of the PFM, not just the abdominal area. This suggests that the pain associated with PD may have a more widespread impact on the pelvic region rather than being localized to the abdomen. Pelvic floor myofascial trigger points (MTrPs) may also exacerbate menstrual pain through the neural pathway.

There is a critical gap in the literature regarding the nature of the association between dysmenorrhea and PFM activity in this population. Yet, it is unknown whether the pain is a cause or result of increased PFM tone, and the nature of the association between menstrual pain and PFM tone in women with PD is also unknown.

So, this study utilizes transabdominal ultrasound (TAU) to examine PFM activity in PD, aiming to clarify how PFM activity contributes to menstrual pain. Understanding these dynamics could lead to preventive strategies and educational efforts highlighting the role of pelvic floor interventions in managing dysmenorrhea, potentially improving treatment methods and overall women's health management.

ELIGIBILITY:
Inclusion Criteria:

* They should be virgin, healthy female physiotherapy students with PD.
* They have regular menstruation (3-8 days in duration, with 21-35 days in between).
* Their ages will range from 18 to 25 years old.
* Their body mass index (BMI) will range from 18 to 24.9 kg/m2.
* Their waist-to-hip ratio will be less than 0.8.

Exclusion Criteria:

* Any urological or gynecological disorders in the previous 12 weeks (e.g., endometriosis, fibroids).
* Fibromyalgia.
* Severe psychiatric or psychological disorders.
* Those who had taken analgesics in the 12 hours before the assessment.
* Abdominal or pelvic surgery within the past six months.

Ages: 19 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Seventy-eight female physiotherapy students with PD will participate in this study. They will be selected randomly from the faculty of physical therapy at Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor muscle (PFM) contraction | 1 month
  Transabdominal ultrasound (TAU) will be used to assess PFM contraction for all females ("cutting off the flow of urine mid-stream") in the three groups.
Pelvic floor muscle (PFM) relaxation | 1 month
  Transabdominal ultrasound (TAU) will be used to assess PFM relaxation during inspiration for all females.

SECONDARY OUTCOMES:
Bladder section of the Australian Pelvic Floor Questionnaire | 1 month
  It will be used to assess the bladder symptoms of pelvic floor dysfunction for all females in the three groups. This section will be scored 0-45, with higher scores meaning more dysfunction
Bowel section of the Australian Pelvic Floor Questionnaire | 1 month
  It will be used to assess the bowel symptoms of pelvic floor dysfunction for all females in the three groups. This section will be scored 0-34, with higher scores meaning more dysfunction
36-Item Short Form Survey Instrument (SF-36) | 1 month
  The SF-36 questionnaire is a self-administered questionnaire containing 36 items. It measures health across eight multi-item dimensions, covering functional status, well-being, and overall health evaluation, each associated with 2-10 possible answers. The response to each question is extrapolated to a standardized set of answers, and the results are transferred to a scale of 0-100, where 0 represents the worst state of health and 100 represents the best state of health measured

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A. Osman, PhD, Study Chair — Assistant Professor; Hossam A. Al Din Hussein Kamel, PhD, Study Director — Professor
Locations (1):
- Cairo University, Giza, Egypt